CLINICAL TRIAL: NCT04754399
Title: Phase 2 Trial of Cannabidiol (CBD) for Treatment of Aromatase Inhibitor-Associated Arthralgias
Brief Title: Cannabidiol (CBD) for Treatment of Aromatase Inhibitor-Associated Arthralgias
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: American Society of Clinical Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: UMCC 2020.041; HUM00182109 (Other: University of Michigan)
Record Dates: First submitted 2021-02-09; First posted 2021-02-15 (Actual); Results first posted 2025-05-09 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Arthralgia; Breast Cancer
Keywords: Cannabidiol
MeSH Terms: conditions — Arthralgia; Breast Neoplasms | interventions — Cannabidiol

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Cannabidiol (CBD) (Experimental): Oral solution given 2x daily.
  Interventions: Drug: Cannabidiol (CBD)

INTERVENTIONS:
Drug: Cannabidiol (CBD) — week 1: 25 mg twice daily, approximately 12 hours apart, with food
  week 2: 50 mg twice daily, approximately 12 hours apart, with food
  week 3: 75 mg twice daily, approximately 12 hours apart, with food
  week 4+: 100 mg twice daily, approximately 12 hours apart, with food
  Other Names: Epidiolex

SUMMARY:
Study of Cannabidol to examine the safety and efficacy of 15 weeks of CBD in postmenopausal women with aromatase inhibitor-associated musculoskeletal symptoms (AIMSS). Investigators are looking to see if patients with joint pain see improvement with the use of CBD.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal according to standard clinical criteria OR receiving concomitant LHRH agonist therapy.
* Taking aromatase inhibitor therapy (anastrozole, exemestane, or letrozole) for adjuvant treatment of breast cancer or for chemoprevention for at least 3 weeks and no more than 2 years at the time of enrollment.
* Planning to take the same AI therapy for at least 15 weeks.
* New or worsening joint pain and/or myalgias since starting the AI therapy.
* Completion of surgery (mastectomy or lumpectomy/partial mastectomy) for treatment of breast cancer at least 3 months prior to enrollment.
* The complete list of inclusion criteria is provided in the protocol.

Exclusion Criteria:

* Metastatic breast cancer.
* Planned surgery during the 15-week study period.
* Clinically significant laboratory abnormalities.
* Use of cannabidiol, THC, or marijuana (oral, inhaled, or topical) within the 6 weeks prior to enrollment.
* History of or currently has suicidal ideation or attempted suicide.
* History of seizure other than febrile seizures in childhood.
* The complete list of exclusion criteria is provided in the protocol.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-04-16 (Actual); Primary Completion 2023-10-10 (Actual); Study Completion 2023-10-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Norah L Henry, MD, PhD, Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Rogel Cancer Center, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fleege NMG, Miller EA, Kidwell KM, Zacharias ZR, Houtman J, Scheu K, Kemmer K, Boehnke KF, Henry NL. Pilot Study of Cannabidiol for Treatment of Aromatase Inhibitor-Associated Musculoskeletal Symptoms in Breast Cancer. Cancer Med. 2025 Aug;14(15):e71117. doi: 10.1002/cam4.71117. PMID 40751295

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1 subject was enrolled but deemed ineligible before starting treatment
Groups:
- Cannabidiol (CBD): Oral solution given 2x daily.
  Cannabidiol (CBD): week 1: 25 mg twice daily, approximately 12 hours apart, with food
  week 2: 50 mg twice daily, approximately 12 hours apart, with food
  week 3: 75 mg twice daily, approximately 12 hours apart, with food
  week 4+: 100 mg twice daily, approximately 12 hours apart, with food
Period: Overall Study
Arm/Group | Cannabidiol (CBD)
Started | 39
Completed | 28
Not Completed | 11
Not completed — Adverse Event | 5
Not completed — Withdrawal by Subject | 6

BASELINE CHARACTERISTICS:
Arm/Group | Cannabidiol (CBD)
Number analyzed (Participants) | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 26
  >=65 years | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 37
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 36
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 39

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change in Brief Pain Inventory (BPI) Worst Pain From Baseline to Week 15
Description: The BPI is a patient self-rating scale that assesses joint pain and stiffness on a scale of 0 (no pain) to 10 (pain as bad as you can imagine). For the purpose of this measure, absolute change for only one BPI item will be assessed, "joint pain and stiffness at its worst in the last week".
Time Frame: Baseline, week 15
Population: 11 patients missing data
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Cannabidiol (CBD)
Number analyzed (Participants) | 28
units on a scale | -2.4 [-3.22 to -1.49]

2. Secondary Outcome: Number of Patients With at Least a 2-point Reduction in BPI Worst Pain From Baseline to Week 15
Description: The BPI is a patient self-rating scale that assesses joint pain and stiffness on a scale of 0 (no pain) to 10 (pain as bad as you can imagine). For the purpose of this measure, change from baseline to week 15 for only one BPI item, "joint pain and stiffness at its worst in the last week", will be assessed.
Time Frame: Baseline, week 15
Population: 11 patients missing data
Measure: Count of Participants; unit: Participants
Arm/Group | Cannabidiol (CBD)
Number analyzed (Participants) | 28
Participants | 17

3. Secondary Outcome: Number of Patients With at Least a 2-point Reduction in BPI Average Pain From Baseline to Week 15
Description: The BPI is a patient self-rating scale that assesses joint pain and stiffness on a scale of 0 (no pain) to 10 (pain as bad as you can imagine). For the purpose of this measure, change from baseline to week 15 for only one BPI item, "joint pain and stiffness on the average", will be assessed.
Time Frame: Baseline, week 15
Population: 11 patients missing data
Measure: Count of Participants; unit: Participants
Arm/Group | Cannabidiol (CBD)
Number analyzed (Participants) | 28
Participants | 14

4. Secondary Outcome: Change in Symptoms From Baseline, as Measured by the PROMIS-29+2 Profile v2.1
Description: The Patient-Reported Outcomes Measurement Information System (PROMIS)-29+2 Profile v2.1 (PROPr) is a validated questionnaire to assess patient-reported symptoms over the past 7 days in 7 PROMIS domains on a scale of 1 (worst) to 5 (best). Raw scores for each domain are calculated and then converted to a T-score, with a mean of 50 and a standard deviation of 10. Higher T-scores represent more of the concept being measured: for fatigue, sleep disturbance, depression, and anxiety, higher scores represent worse symptoms; for physical functioning, ability to participate in social roles and activities, and cognitive function-abilities, higher scores mean better function.
Time Frame: Baseline, week 15
Population: 11 patients missing data
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cannabidiol (CBD)
Number analyzed (Participants) | 28
score on a scale
  Pain interference | -6.5 (7.2)
  Pain intensity | -1.9 (2.1)
  Cognitive function | 2.0 (1.2)
  Depression | -1.7 (4.5)
  Ability to participate in social roles/activities | 5.7 (8.0)
  Anxiety | -3.4 (6.0)
  Physical function | 3.9 (5.3)
  Fatigue | -3.3 (6.9)
  Sleep disturbance | -3.7 (6.6)

5. Secondary Outcome: Number of Treatment Related Adverse Events
Description: Treatment related adverse events include those that are determined to be possibly, probably or definitely related to the study drug. Number of events will be reported by dose level and grade, per Common Terminology Criteria for Adverse Events (CTCAE) v.5.
Time Frame: End of study (15 weeks)
Measure: Number; unit: number of events
Arm/Group | Cannabidiol (CBD)
Number analyzed (Participants) | 39
number of events
  Agitation- grade 2- 25mg BID dose | 1
  Nausea- grade 1- 25mg BID dose | 1
  Flushing- grade 1- 25mg BID dose | 1
  Anxiety- grade 1- 50mg BID dose | 1
  Rash- grade 2- 50mg BID dose | 2
  Nausea- grade 1- 50mg BID dose | 1
  Depression- grade 1- 75 mg BID dose | 1
  Stomach Pain- grade 1- 75 mg BID dose | 1
  Fatigue- grade 1- 75 mg BID dose | 1
  Headache- grade 1- 75 mg BID dose | 1
  Hyponatremia- grade 1- 75 mg BID dose | 1
  Hyperglycemia- grade 1- 75 mg BID dose | 1
  Peripheral motor neuropathy- grade 1- 100 mg BID dose | 1
  Peripheral motor neuropathy- grade 2- 100 mg BID dose | 1
  Fatigue- grade 1- 100 mg BID dose | 1
  Memory impairment- grade 1- 100 mg BID dose | 1
  Anorexia- grade 2- 100 mg BID dose | 1
  Diarrhea- grade 2- 100 mg BID dose | 1
  Nausea- grade 1 - 100 mg BID dose | 2
  alanine aminotransferase increased- grade 1- 100 mg BID dose | 1
  Oral Pain- grade 1- 100 mg BID dose | 1
  Gastroesophageal reflux disease- grade1- 100 mg BID dose | 1
  Increased creatinine- grade 1- 100 mg BID dose | 1
  stomach pain- grade 1- 100 mg BID dose | 1
  dizziness- grade 1- 100 mg BID dose | 1
  Headache- grade 1- 100 mg BID dose | 1

6. Secondary Outcome: Number of Participants With Undetectable Levels of Estradiol
Description: The number of participants with undetectable levels of estradiol circulating in blood plasma will be reported at baseline and 15 weeks.
Time Frame: Baseline and week 15
Population: All enrolled patients would be analyzed; however, 3 samples are missing for baseline and 9 for week 15
Measure: Count of Participants; unit: Participants
Arm/Group | Cannabidiol (CBD)
Number analyzed (Participants) | 36
Participants
  Baseline | 8
  15 Weeks: number analyzed (Participants) | 30
  15 Weeks | 4

ADVERSE EVENTS:
Time Frame: All adverse event data (serious and non-serious) collected from the time of the initial study treatment administration through 30 days after the last dose of study treatment. Up to 2 years.
Groups:
- Cannabidiol (CBD)- Week 1: Oral solution given 2x daily.
  Cannabidiol (CBD): week 1: 25 mg twice daily, approximately 12 hours apart, with food
- CBD- Week 2: Oral solution given 2x daily.
  Cannabidiol (CBD):
  week 2: 50 mg twice daily, approximately 12 hours apart, with food
- CBD- Week 3: Oral solution given 2x daily.
  Cannabidiol (CBD):
  week 3: 75 mg twice daily, approximately 12 hours apart, with food
- CBD- Week 4: Oral solution given 2x daily.
  Cannabidiol (CBD):
  week 4+: 100 mg twice daily, approximately 12 hours apart, with food
Arm/Group | Cannabidiol (CBD)- Week 1 | CBD- Week 2 | CBD- Week 3 | CBD- Week 4
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/39 | 0/39 | 0/39
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/39 | 0/39 | 0/39
Other Adverse Events (participants affected / at risk) | 12/39 | 3/39 | 8/39 | 11/39
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cannabidiol (CBD)- Week 1 (N=39) | CBD- Week 2 (N=39) | CBD- Week 3 (N=39) | CBD- Week 4 (N=39)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bladder infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Creatinine increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Flushing (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (2) | 0 (0) | 1 (2) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (4) | 0 (0) | 0 (0) | 2 (3)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Stomach pain (Gastrointestinal disorders) | 1 (2) | 0 (0) | 1 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-07-20): https://cdn.clinicaltrials.gov/large-docs/99/NCT04754399/Prot_SAP_002.pdf
  • Informed Consent Form (2022-08-31): https://cdn.clinicaltrials.gov/large-docs/99/NCT04754399/ICF_001.pdf